CLINICAL TRIAL: NCT00289445
Title: Open, Multi-center Phase I/II Trial With Mitomycin C in Combination With 5-Fluorouracil and Folinic Acid in Pretreated Patients With Metastatic Gastrointestinal Cancer
Brief Title: Study With Mitomycin c/5-FU/FA in Pretreated Gastrointestinal Cancer Patients With Metastases (>= Second-line Treatment)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jth_003
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Gastrointestinal Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasm Metastasis | interventions — Mitomycin; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: Mitomycin C
Drug: 5-FU
Drug: Folinic acid

SUMMARY:
The aim of this study was to define the maximum tolerated dose (MTD) of bolus mitomycin C (MMC) in combination with 24 h-continuous infusion of 5-fluorouracil (FU) plus folinic acid, and to assess the toxicity and activity in patients with previously treated colorectal and gastric cancer. Escalating doses of MMC starting from 6 mg m(-2) in 2 mg m(-2)-steps to a maximum of 10 mg m(-2) were applied on days 1 and 22, given to fixed doses of 5-FU (2.600 mg m(-2)) as 24 h infusion and folinic acid 500 mg m(-2) prior to 5-FU weekly for 6 weeks

ELIGIBILITY:
Inclusion Criteria:

Phase 1 (dose escalation)

* patients with histological proven gastrointestinal neoplasms, without standard therapy option
* measurable or evaluable disease
* >= second-line therapy (metastasized stage) Phase 2 (efficacy)
* patients with proven colorectal neoplasms
* measurable disease, metastasized
* previous chemotherapy with 5-FU/FA ("AIO-regimen")
* age between 18 and 75 years, both male and female
* life expectancy > 3 months
* WHO-performance status <= 2
* adequate bone marrow function: hemoglobin >= 10 mg/dl, neutrophils >= 2.0 * 1000000000/l, thrombocytes >= 150 * 1000000000/l
* adequate renal and liver function: bilirubin <= 1.25 * ULN(<= 1.5 ULN * by liver metastases), creatinine <= 1.25 * ULN, ASAT and ALAT <= 3 * ULN (<= 5* ULN by liver metastases; AP <= 3* ULN
* written informed consent prior to inclusion into the study

Exclusion Criteria:

* pretreated with mitomycin c
* contraindication concerning 5-FU (e.g. anxiety, myocardial infarction within last 6 months, significant toxicities during previous therapy with 5-FU
* florid infections
* ileus or subileus, morbus crohn or colitis, ulcerative
* actual chronic diarrhea
* other uncontrolled severe concurrent disease excluding cytotoxic intervention
* second malignancy except basal cell carcinoma or cervical carcinoma in situ
* known cns metastases or carcinomatous leptomeningitis
* pregnancy or lactation period
* no effective contraception
* concomitant treatment with another antineoplastic agents
* participation in another clinical trial within the last 4 weeks
* patients being unwilling or unable to undergo trial specific procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) of bolus mitomycin C (MMC) in combination with 24 h-continuous infusion of 5-fluorouracil (FU) plus folinic acid
toxicity
activity

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bokemeyer, MD, Principal Investigator — University Hospital Tuebingen (PI until 30Nov2004); Joerg T Hartmann, MD, Principal Investigator — University Hospital Tuebingen